CLINICAL TRIAL: NCT02235181
Title: An Open Randomised Trial of the Arabin Pessary to Prevent Pre-term Birth in Twin Pregnancy in Woman With a Short Cervix (STOPPIT-2)
Brief Title: An Open Randomised Trial of the Arabin Pessary to Prevent Pre-term Birth in Twin Pregnancy
Acronym: STOPPIT-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STOPPIT-2
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Twin Pregnancy With Antenatal Problem
Keywords: Twin Pregnancy; Prevention of Preterm birth; Short Cervix; Arabin cervical pessary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Treatment (No Intervention): Women will be allocated to standard treatment, currently this is no treatment.
- Arabin pessary (Active Comparator): The Arabin cervical pessary will be inserted between 18 and 20+6 days gestation and removed between 35 and 36+6 weeks gestation unless Labour occurs sooner.
  Interventions: Device: Arabin Cervical Pessary

INTERVENTIONS:
Device: Arabin Cervical Pessary — The Arabin pessary is CE-certified for preventing Spontaneous Preterm Birth (SPB) (CE 0482 / EN ISO 13485: 2003 annex III of the council directive 93/42 EEC) and is being used in this study as per the CE certification and manufacturer's guidance.
  Arms: Arabin pessary

SUMMARY:
This study aims to determine whether the Arabin cervical pessary prevents preterm birth in women with a twin pregnancy and a short cervix.

DETAILED DESCRIPTION:
STOPPIT-2 is a multicentre open label randomised controlled trial of the Arabin pessary (CE marked Device) versus Standard treatment in women with twin pregnancy. The study is in two phases - a SCREENING phase, in which women with a short cervix (cervical length of ( less or equal to 35mm) will be identified, and a TREATMENT phase, in which women with a short cervix will be randomised to treatment with Arabin pessary or Standard treatment. Women will be seen in the antenatal clinic setting.

An internal pilot phase will take place, with ten interviews being conducted with pregnant women to explore the acceptability of proposed methods of recruitment, their information requirements, their views of the consent and randomisation processes, and the delivery of the intervention, including the screening component. The interviews will also explore their understanding and expectations of trial participation. The findings of this pilot phase will feed into the next phase of the trial and support the design of the interview guides for the main nested qualitative study.

This pilot phase is separate from the main study. Later on we will ask both women and healthcare professionals about their experiences of the study, via questionnaires and face-to-face interviews.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting with twin pregnancy (monochorionic or dichorionic)
* Women with gestation established by scan at ≤16 weeks according to NICE guidelines.
* Women aged 16 years or older
* Women wishing to participate in both the SCREENING and RANDOMISATION phase of the study

Exclusion Criteria:

* Women unable to give written informed consent
* Women with known significant congenital structural or chromosomal fetal anomaly at the time of inclusion
* Women with existing or planned cervical cerclage in the current pregnancy
* Women who with existing or planned (prior to 20+6 weeks gestation) treatment for twin to twin transfusion syndrome in the current pregnancy
* Women with suspected or proven rupture of the fetal membranes at the time of recruitment
* Women with singleton pregnancy or higher order multiple pregnancies
* Women with known sensitivity, contraindication or intolerance to silicone
* Women involved in a clinical trial of an investigational medicinal product (CTIMP)

Ages: 16 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2228 (Actual)
Dates: Start 2014-11-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
The Arabin cervical pessary reduces spontaneous preterm labour leading to preterm birth | Delivery of the babies
  Gestation at delivery
Neonatal Outcomes | within 4 weeks after expected date of delivery
  The investigators will collect a number of measures to ascertain neonatal well being.

SECONDARY OUTCOMES:
The profile of cervical length measurements in women with twin pregnancy in the UK | 18-20 weeks gestation
  Cervical length
Participant Satisfaction | 36 weeks gestation
  Acceptability questionnaire
Health economics | 18-20 weeks gestation until 4 weeks postnatal
  cumulative hospital costs

CONTACTS AND LOCATIONS:
Overall Officials: Jane E Norman, MD, Principal Investigator — University of Edinburgh
Locations (57):
- UZ Leuven, Leuven, Belgium
- United Kingdom (56):
  - Countess of Chester, Chester, Cheshire
  - St Mary's Hospital, Manchester, Cheshire
  - Chesterfield Royal Hospital, Chesterfield, Derbyshire
  - Derriford Hospital, Plymouth, Devon
  - Poole Hospital, Poole, Dorset
  - Basildon hospital, Basildon, Essex
  - Hillingdon Hospital, Uxbridge, Greater London
  - Royal Bolton Hospital, Bolton, Lancashire
  - Royal Preston Hospital, Preston, Lancashire
  - Croydon hospital, Croydon, London
  - Simpson Centre for Reproductive Health, Royal Infirmary Hospital, Edinburgh, Edinburgh, Lothian
  - Pinderfields Hospital, Wakefield, Mid Yorkshire
  - Royal Victoria Hospital, Newcastle upon Tyne, North East
  - Wansbeck General Hospital, Ashington, Northumbria
  - North Tyneside General Hospital, North Shields, Northumbria
  - St Helier Hospital, Carshalton, Surrey
  - Epsom Hospital, Epsom, Surrey
  - George Eliot, Nuneaton, Warwickshire
  - Birmingham Womens Hospital, Birmingham, West Midlands
  - Russells Hall Hospital, Dudley, West Midlands
  - Bradford Royal Infirmary, Bradford, Yorkshire
  - Leeds University Hospital Trust, Leeds, Yorkshire
  - Aberdeen Maternity Hospital, Aberdeen
  - Birmingham Heartlands Hospital, Birmingham
  - Lancashire Women's and Newborn Centre, Burnley
  - Rosie Maternity Hospital, Cambridge
  - Leighton Hospital, Crewe
  - Royal Devon & Exeter, Exeter
  - Queen Elizabeth Hospital, Gateshead
  - Princess Royal Maternity Hospital, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Arrowe Park Hospital, Wirral, Liverpool
  - Liverpool Women's Hospital, Liverpool
  - Whiston Hospital, Liverpool
  - St Johns Hospital, Livingston
  - Homerton University Hospital NHS Foundation Trust, London
  - Newham Hospital, London
  - Queen Charlottes' Hospital, London
  - Royal London Hospital, London
  - St Georges Hospital, London
  - St Thomas Hospital, London
  - St. Mary's, London
  - University College Hospital, London
  - Whipps Cross Hospital, London
  - James Cook Hospital, Middlesbrough
  - Norfolk and Norwich Hospital, Norwich
  - City Hospital NUH NHS Trust, Nottingham
  - Queens Medical Centre, NUH NHS Trust, Nottingham
  - Salisbury District Hospital, Salisbury
  - Jessop Wing, Sheffield Teaching Hospitals NHS FT, Sheffield
  - Princess Anne Hospital, Southampton
  - Royal Stoke University Hospital University Hospitals of North Midlands, Stoke
  - Sunderland Royal Hospital, Sunderland
  - Royal Cornwall, Truro
  - New Cross Hospital, Wolverhampton
  - Wrexham Maelor, Wrexham

IPD SHARING:
Plan to Share IPD: Yes
to be confirmed

REFERENCES:
- [Derived] Norman JE, Norrie J, MacLennan G, Cooper D, Whyte S, Chowdhry S, Cunningham-Burley S, Neilson AR, Mei XW, Smith JB, Shennan A, Robson SC, Thornton S, Kilby MD, Marlow N, Stock SJ, Bennett PR, Denton J. The Arabin pessary to prevent preterm birth in women with a twin pregnancy and a short cervix: the STOPPIT 2 RCT. Health Technol Assess. 2021 Jul;25(44):1-66. doi: 10.3310/hta25440. PMID 34219633
- [Derived] Norman JE, Norrie J, MacLennan G, Cooper D, Whyte S, Chowdhry S, Cunningham-Burley S, Mei XW, Smith JBE, Shennan A, Robson SC, Thornton S, Kilby MD, Marlow N, Stock SJ, Bennett PR, Denton J; STOPPIT-2 collaborative group. Evaluation of the Arabin cervical pessary for prevention of preterm birth in women with a twin pregnancy and short cervix (STOPPIT-2): An open-label randomised trial and updated meta-analysis. PLoS Med. 2021 Mar 29;18(3):e1003506. doi: 10.1371/journal.pmed.1003506. eCollection 2021 Mar. PMID 33780463
- [Derived] Norman JE, Norrie J, Maclennan G, Cooper D, Whyte S, Cunningham Burley S, Smith JBE, Shennan A, Robson SC, Thornton S, Kilby MD, Marlow N, Stock SJ, Bennett PR, Denton J. Open randomised trial of the (Arabin) pessary to prevent preterm birth in twin pregnancy with health economics and acceptability: STOPPIT-2-a study protocol. BMJ Open. 2018 Dec 6;8(12):e026430. doi: 10.1136/bmjopen-2018-026430. PMID 30530477
- See also: STOPPIT2 Study page — https://w3.abdn.ac.uk/hsru/STOPPIT2/